CLINICAL TRIAL: NCT02329340
Title: Safety Skills Training: Parents of School-Aged Children
Acronym: SAS_2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Susan Schroeder, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBIR76R-2; R44HD048005 (NIH)
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Injuries
Keywords: child safety; injury; prevention; computer; internet
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Am Academy of Pediatrics print materials (Active Comparator): In-person session to read online version of American Academy of Pediatrics The Injury Prevention Program (TIPP sheets) childhood injury prevention print materials, followed by access to the TIPP sheets for 30 days.
  Interventions: Behavioral: Am Academy of Pediatrics print materials
- Family Safety 1-2-3 (Experimental): In-person session to view video and text-based interactive web site on injury prevention information and strategies, followed by 8 emails delivered over a 30-day period inviting participant to view additional child safety videos.
  Interventions: Behavioral: Family safety 1-2-3

INTERVENTIONS:
Behavioral: Am Academy of Pediatrics print materials — Print materials of injury prevention content.
  Other Names: The Injury Prevention Program; tip sheets
  Arms: Am Academy of Pediatrics print materials
Behavioral: Family safety 1-2-3 — Theoretically based school-aged childhood injury prevention videos for families
  Arms: Family Safety 1-2-3

SUMMARY:
Injuries are the leading cause of death and disability in children in America. Most injuries can be prevented when parents implement effective child safety practices. This project will create a behaviorally based program to teach parents what to do to prevent injuries to their school aged child, in an effort to reduce the number of injuries, hospitalizations, medical costs, and missed work days.

DETAILED DESCRIPTION:
This project will produce a comprehensive, interactive multimedia (IMM) program to teach childhood injury prevention skills to parents of children 6 through 11 years of age. This is one of a four-part series of funded programs to address injury prevention issues for three age groups of children (birth through 24 months, 2-5 years of age and 6-11 years of age). The program will be created in three formats: Internet/intranet, CD-ROM, and linear video (DVD) suitable for use in homes, worksites, medical settings, service agencies, and health information Web sites. On-screen narrators will guide the user through program material comprised of short video presentations, modeling vignettes demonstrating desired behaviors, supportive testimonials, and suggestions for modifications to home and recreational environments.

ELIGIBILITY:
Inclusion Criteria:

* The basic lower age limit for parents or guardians of children aged 6-11 for this study was 18. Parents or legal guardians could potentially be as old as 65 or older.

Exclusion Criteria:

* Only English-speaking participants were accepted because the program was developed only for English speakers. All English-speaking parents or guardians living in the U.S., with children aged 6-11 years old, who wished to participate were included. Parents under 18 were excluded from this online study because parental consent cannot be obtained online.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Behavioral measure: identification of correct/incorrect car booster safety seat, seat belt, and bicycle helmet placement | Immediate posttest and 30-day follow-up
  Parents viewed 2 car seat installations and were asked whether 7 car booster safety seat situations (e.g., age of the child for the seat) and 7 seat belt installations (e.g., placement of the seat belt) were correct or incorrect. Parents also viewed a bicycle helmet on a dummy and were asked to identify whether 2 helmet situations were correct or incorrect.

SECONDARY OUTCOMES:
Knowledge of injury prevention strategies | immediate posttest and 30-day follow-up
  An injury prevention knowledge scale was created across all content areas. The injury prevention knowledge scale contained 39 items (e.g., "To prevent scald injuries, hot water heaters should be set to …") for all age groups. The injury prevention knowledge scale represented the percent of items correctly endorsed.
Attitudes and beliefs about injury prevention strategies | immediate posttest and 30-day follow-up
  An injury prevention attitudes & beliefs scale was created across all content areas (e.g., "A family emergency plan is extremely important strategy to keep your family safe in case of a fire."). Twenty-five items assessed attitudes & beliefs for the 6-9 year age group and 24-items the 10-11 age group (alpha = .81 for both younger and older children). All items were assessed using a 5-point Likert scale with 1 = strongly disagree to 5 = strongly agree.
Self-efficacy for engaging in injury prevention strategies | immediate posttest and 30-day follow-up
  An injury prevention self-efficacy scale was created from 29 items across all content areas for all age groups (e.g., "How confident are you that you know how to test the temperature of your water heater?") (alpha = .91 for all age groups) All items were assessed using a 5-point Likert scale with 1 = strongly disagree to 5 = strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne H Grilley Swartz, MPH, CHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States